CLINICAL TRIAL: NCT02266979
Title: Study to Determine Appropriate Nurse: Patient Ratios in Peritoneal Dialysis Programs
Status: Completed | Type: Observational
Sponsor: Ana Elizabeth Prado Lima Figueiredo (Other)
Responsible Party: Sponsor-Investigator, Ana Elizabeth Prado Lima Figueiredo, Professor, Pontificia Universidade Católica do Rio Grande do Sul
Organization: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Other Study IDs: AEFIIRPDstaff2014
Record Dates: First submitted 2014-09-28; First posted 2014-10-17 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Renal Failure
Keywords: peritoneal dialysis; nursing staff; nursing activities; Personnel Downsizing
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
As the resolution of the Brazilian Federal Council of Nursing (COFEN) sizing the framework of nursing professionals is essential to ensure the safety and quality of patient care. To achieve such goals actions are needed to evaluate the variety of tasks and performance specific to each area in nursing profession. The National Agency for Health Surveillance (ANVISA), through Board Resolution (RDC-154) determines that the nurse to patient ratio is 1 to 30 in hemodialysis and 1 to 50 on peritoneal dialysis, however these targets are not based on any evidence, and same apply to other Latin-American countries. Objective: To determine the appropriate nurse: patient ratio for peritoneal dialysis unit. Method: This research will be developed in two phases. The first with an observational design with descriptive and qualitative approach. There will be a focus group with experts in the field, to defined the activities and responsibilities of the peritoneal dialysis nurse, and produce a tool with a list of activities. A time-orientated score will be created. In the second stage a cross-sectional quantitative approach will be used. To apply the instrument from by direct observation of activities performed by nurses during their workday. With the instrument activities will be timed and the overall time of each nursing activity will be determined by multiplying the time spent by the total number of patients. It is expected tat this strategy will increase time on treatment and/or decrease dropout rates, by developing an easy test/ formula application to determine the correct ratio according to the peritoneal dialysis program. This tool will provide better outcomes for patients as well as allow for growth of peritoneal dialysis programs with qualified assistance and patient safety.

DETAILED DESCRIPTION:
Research question:

Can a time-oriented score system and expert consensus be applied to PD to develop an easy and repeatable system to evaluate work load for peritoneal dialysis nurses to achieve the best outcomes and allow for planned growth of the unit?

ELIGIBILITY:
Inclusion Criteria:

* To have at least one year of experience with peritoneal dialysis

Exclusion Criteria:

* Not applicable
* Consent withdraw

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Renal nurses, master and PhD nurse experts in peritoneal dialysis to develop a list of activities to be timed
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
number of activities ( direct or indirect care) performed by peritoneal dialysis nurse | 6 months
  after focal groups a list we all activities performed by PD nurses will be prepared

SECONDARY OUTCOMES:
time to perform activities | 6 months
  the time spend to perform each activities will be measured to calculate time spent with patients

CONTACTS AND LOCATIONS:
Overall Officials: Ana E Figueiredo, RN, PhD, Principal Investigator — Pontificia Universidade Católica do Rio Grande do Sul
Locations (1):
- Pontificia Universidade Católica Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil